CLINICAL TRIAL: NCT02108236
Title: Effectiveness and Safety of Acupuncture for Obesity and Over-weight People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wang Ling Shu, the head of institute of chinese medicine and translational science of First Affiliated Hospital, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acupuncture-Obesity-2014-3
Record Dates: First submitted 2014-03-30; First posted 2014-04-09 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Overweight
Keywords: acupuncture; chinese traditional medicine
MeSH Terms: conditions — Obesity; Overweight | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blank control group (No Intervention): A control group of patients is put on a waiting list for no intervention and remaining unchanged lifestyle.
- intervention group (Active Comparator): An intervention group of patients is put on a waiting list for acupuncture treatment.
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — Zhong-wan (RN12), Liang-men (ST21), Shui-fen (RN9) and Qi-hai (RN6) and bilateral acupuncture points Dai-mai (GB26), Tian-shu (ST25), Zu-sanli (ST36), Feng-long(ST40) and Liang-qiu(ST34) will be applied through the skin by acupuncture for 30 minutes every time. Electro-acupuncture apparatus will be connected to both Dai-mai, Zu-sanli and Feng-long, Zhong-wan and Qi-hai for 30 minutes with interrupted waves (2/100HZ).
  Arms: intervention group

SUMMARY:
To determine the efficacy and safety of acupuncture for obesity and overweight people in China.

ELIGIBILITY:
Inclusion Criteria:

* The individuals is phlegm-dampness constitution and female.
* Age is between 18 and 45 years.
* BMI is between 24 and 50.
* The individuals voluntarily sign the informed consent form.
* The individuals live in Harbin City of China.

Exclusion Criteria:

* Secondary obesity, eg:pituitary diseases, hypothalamic disorder, hypothyroidism, pancreatic diseases，hyperadrenocorticism, postmenopausal obesity etc.
* The individuals with server cardiovascular and cerebrovascular diseases and cancer.
* Having therapy for obesity in the last three months.
* The individuals do not adhere to the treatment or are with other treatments.
* Female individuals with pregnancy, lactation and planning a pregnancy in the two months.
* Critical patients or patients combined with liver and kidney damage.
* Individuals with visual and auditory memory disorders or psychosis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
body mass index(BMI) | 2 month after treatment

SECONDARY OUTCOMES:
waist-to-hip ratio (WHR) | 2 month after treatment
Blood sugar | 2 month after treatment
Total cholesterol | 2 month after treatment
Triglycerides | 2 month after treatment
High-density lipoprotein cholesterol | 2 month after treatment
Low-density lipoprotein cholesterol | 2 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sun Zhongren, Principal Investigator — First Affiliated Hospital of Heilongjiang Chinese Medicine University
Locations (1):
- The First Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang, China